CLINICAL TRIAL: NCT04629534
Title: Mothers' Own Milk Optimization for Preterm Infants Project (MoMO PIP): Maternal Diet and Vitamin D Supplementation Effects on Preterm Infants, a Randomized Control Pilot Study.
Brief Title: Mothers' Own Milk Optimization for Preterm Infants Project (MoMO PIP) Pilot Study
Acronym: MoMO PIP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment, lack of funding
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Raechel Irons, Neonatal-Perinatal Fellow, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00099911
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Vitamin D Deficiency; Nutritional Deficiency
Keywords: Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Malnutrition | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: High dose Cholecalciferol
- Group B (Placebo Comparator)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: High dose Cholecalciferol — Mothers in experimental group will receive 6,000 IU of vitamin D in addition to their prenatal vitamin, daily for 3 months. Infants in this group will receive placebo vitamin D drops
  Other Names: 6,600 IU of cholecalciferol
  Arms: Group A
Drug: Cholecalciferol — Mothers in placebo control group will receive 600 IU of vitamin D in the form of their prenatal vitamin along with placebo vitamin D. Infants of the mothers in this group will receive standard 400 IU of vitamin D
  Other Names: 600 IU of cholecalciferol
  Arms: Group B

SUMMARY:
The overall goal of this study is to assess maternal vitamin D status along with diet, and milk composition, and in turn, to evaluate if infant vitamin D status can be improved with increased maternal supplementation and diet education. The central hypothesis is that by maximizing maternal vitamin D status in breastfed, preterm infants (<35 weeks), there will be an increase infant 25(OH)D status at 1,2, and 3 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Women with documentation of fully breastfeeding who present within one month of delivery, who are 18-45 years old and in good general health will be eligible for participation.
* Infants <35 weeks corrected gestational age at birth

Exclusion Criteria:

* NO DMI/DMII, HTN, or parathyroid disease IF thyroid issues, currently euthyroid
* Multiple gestations
* No liver disease
* No major congenital abnormalities
* No kidney disease
* No inborn errors of metabolism
* No parathyroid disease
* No disorders of calcium metabolism
* No antiepileptics
* No steroids
* No congenital heart disease
* No severe illness at birth deemed incompatible with survival

Ages: 0 Days to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raechel Irons, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Shawn Jenkins Childrens Hospital, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study contained dyads of mother's and their newborn infants. Double-blinded control randomized study
Pre-assignment Details: This study involves mother and infant dyads. There were 8 individual participants enrolled onto the study. 4 mothers and 4 infants which is equivalent to 4 dyads. Group A had 2 dyads (4 individual participants). Group B also had 2 dyads (4 individual participants) However, if an infant became ineligible but mother still qualified, she could remain in the study separately. The participant flow reflects the individual participants.
Groups:
- Group A: High dose Cholecalciferol: Mothers in experimental group will receive 6,000 IU of vitamin D in addition to their prenatal vitamin, daily for 3 months. Infants of these mothers will receive placebo drops.
- Group B: Cholecalciferol: Mothers in placebo control group will receive 600 IU of vitamin D in the form of their prenatal vitamin along with placebo vitamin D. Infants of these mothers will receive standard 400 IU of vitamin D drops.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 4 | 4
Completed | 3 (An infant with withdrawal as they became ineligible due to physician discretion.) | 2 (A mother and infant dyad were removed as she stopped breast feeding and no longer met qualifications for this study)
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Mother/Infant Dyads that delivered at the Medical University of South Carolina between 24-34 weeks gestation were eligible for enrollment. Mother's and infants are counted separately in these results as 1 mother continued the study after her child was removed for parental preferences.
Groups:
- Group A: High dose Cholecalciferol: Mothers in experimental group will receive 6,000 IU of vitamin D in addition to their prenatal vitamin, daily for 3 months.
- Group B: Cholecalciferol: Mothers in placebo control group will receive 600 IU of vitamin D in the form of their prenatal vitamin along with placebo vitamin D.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] — Population: Means reflect only mother's ages
  years
    Mothers: number analyzed (Participants) | 2 | 2 | 4
    Mothers | 28.5 [26 to 31] | 24.5 [23 to 26] | 27 [23 to 31]
Age, Customized [Mean (Full Range); unit: weeks] — Corrected Gestational Age (CGA) of infants enrolled in the study. Population: moms are measured in years and baby's are measured in weeks of age at birth
  weeks
    Infants: number analyzed (Participants) | 2 | 2 | 4
    Infants | 28.5 [26 to 31] | 30 [28 to 32] | 29.25 [26 to 32]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For analyzing this population I separated out mothers and infants.
  Participants
    Mothers: number analyzed (Participants) | 2 | 2 | 4
    Mothers: Female | 2 | 2 | 4
    Mothers: Male | 0 | 0 | 0
    Infants: number analyzed (Participants) | 2 | 2 | 4
    Infants: Female | 1 | 1 | 2
    Infants: Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Mothers and infants were analyzed separately
  Participants
    Mothers: number analyzed (Participants) | 2 | 2 | 4
    Mothers: American Indian or Alaska Native | 0 | 0 | 0
    Mothers: Asian | 0 | 0 | 0
    Mothers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Mothers: Black or African American | 1 | 1 | 2
    Mothers: White | 1 | 1 | 2
    Mothers: More than one race | 0 | 0 | 0
    Mothers: Unknown or Not Reported | 0 | 0 | 0
    Infants: number analyzed (Participants) | 2 | 2 | 4
    Infants: American Indian or Alaska Native | 0 | 0 | 0
    Infants: Asian | 0 | 0 | 0
    Infants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Infants: Black or African American | 1 | 1 | 2
    Infants: White | 1 | 1 | 2
    Infants: More than one race | 0 | 0 | 0
    Infants: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Though these are mother/infant dyads. All participants are reported individually.
  participants
    United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants With Sufficient 25(OH)D Stores at 3 Months
Description: Number of infants with 25(OH)D levels > 20 ng/mL
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

2. Primary Outcome: Number of Mothers With Sufficient 25(OH)D Stores at 3 Months
Description: Number of mothers with 25(OH)D levels >20 ng/mL
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 1 | 1

3. Primary Outcome: Number of Mothers With Elevated Calcium Concentrations at 1 Month
Description: Number of mothers with serum calcium > 10.5 mg/dL
Time Frame: 1 month post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

4. Primary Outcome: Number of Mothers With Elevated Calcium Concentrations at Month 2
Description: Number of mothers with serum calcium > 10.5 mg/dL
Time Frame: 2 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

5. Primary Outcome: Number of Mothers With Elevated Calcium Concentrations at Month 3
Description: Number of mothers with serum calcium > 10.5 mg/dL
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

6. Primary Outcome: Number of Mothers With Elevated Urine Calcium Creatinine Ratio at Month 1
Description: Number of mothers with serum calcium > 1.0 mmol/mmol
Time Frame: 1 month post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

7. Primary Outcome: Number of Mothers With Elevated Urine Calcium Creatinine Ratio at Month 2
Description: Number of mothers with urine calcium/creatinine ratio > 1.0 mmol/mmol
Time Frame: 2 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

8. Primary Outcome: Number of Mothers With Elevated Urine Calcium Creatinine Ratio at Month 3
Description: Number of mothers with urine calcium/creatinine ratio > 1.0 mmol/mmol
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

9. Primary Outcome: Number of Infants With Elevated Calcium Concentration at Month 1
Description: Number of infants with serum calcium > 11.0 mg/dL
Time Frame: 1 month post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

10. Primary Outcome: Number of Infants With Elevated Calcium Concentration at Month 2
Description: Number of infants with serum calcium > 11.0 mg/dL
Time Frame: 2 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

11. Primary Outcome: Number of Infants With Elevated Calcium Concentration at Month 3
Description: Number of infants with serum calcium > 11.0 mg/dL
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Data was collected over a 3 month period.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to a small number of subjects analyzed with difficulty in enrollment. Technical issue with calculating total vitamin D intake through formula fortification and TPN along with the study drugs which can skew our data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT04629534/Prot_002.pdf